CLINICAL TRIAL: NCT06055712
Title: Antibiotic Prophylaxis in Pediatric Open Fractures
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Raju Sivashanmugam, Associate Professor, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 30873
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Fractures, Open; Infections
Keywords: Pediatric open fracture; Antibiotic regimen; Infection rate
MeSH Terms: conditions — Fractures, Open; Infections | interventions — Cefazolin; Cephalexin

STUDY DESIGN:
Intervention Model Description: This is a prospective clinical trial in which patients will be assigned a study arm in sequential fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- One dose of IV cefazolin (Active Comparator): Patients in group A will receive one dose of IV cefazolin and will have no further antibiotic administration.
  Interventions: Drug: Cefazolin
- 24 hours IV cefazolin (Active Comparator): Patients in group B will receive a dose of IV cefazolin every 8 hours for 24 hours (a total of 3 doses).
  Interventions: Drug: Cefazolin
- 24 hours IV cefazolin plus 5 days oral cephalexin (Active Comparator): Patients in group C will receive a dose of IV cefazolin every 8 hours for 24 hours (a total of 3 doses). Additionally, they will be instructed to take 5 days of oral cephalexin.
  Interventions: Drug: Cefazolin; Drug: Cephalexin

INTERVENTIONS:
Drug: Cefazolin — Intravenous dose(s).
Drug: Cephalexin — Five days oral.
  Arms: 24 hours IV cefazolin plus 5 days oral cephalexin

SUMMARY:
This research will involve a prospective study on infection rates after grade 1 or 2 open fractures in the skeletally immature pediatric population. There will be 3 arms: one dose intravenous cefazolin, 24 hours intravenous cefazolin, and 24 hours intravenous cefazolin plus 5 days of oral cephalexin.

DETAILED DESCRIPTION:
Pediatric patients presenting with open fractures will be screened for eligibility at the time of presentation. Informed consent form discussion will take place within 8 hours of the patient's presentation, or before their second dose of antibiotics would be due (if randomized to group 2 or 3).

Upon arrival to the ED with an open fracture (grade I or II), the patient is assessed and care is initiated based on patient presentation. Patients are given an IV for medication administration and receive the first dose of antibiotics (cefazolin) as soon as possible. This is standard of care.

Treatment of the fracture includes irrigation with saline (at least 1 liter depending on wound size). The fracture then needs to be stabilized and wound closed. Patients are taken to the trauma room typically within 8 hours of presentation for sedation and closed reduction of the fracture. These practices are standard of care.

If the patient and guardian consent to the study, the patient will be randomized to one of three study arms:

A) one dose of IV cefazolin B) 24 hours IV cefazolin (3 doses Q8hrs) C) 24 hours IV cefazolin (3 doses Q8hrs) plus 5 days oral cephalexin.

Patients in group A will have no further antibiotic administration, assuming they received their first (and only) dose as soon as possible upon arrival. Patients in groups B and C will need to receive their second doses of IV cefazolin 8 hours after administration of the first dose. This is why we plan to consent the patients/guardians within 8 hours of presentation.

Aside from antibiotic administration, all other treatment will be standard of care. Patients will undergo closed reduction and any other medical management deemed necessary. Prior to discharge, participants will be educated on how to identify symptoms of infection. It is standard of care to discuss this during discharge education.

Frequency of follow up will be determined by standard of care treatment plan for age and fracture type. This is at the discretion of the physician. Typical follow up is at 1 week then 1 or 2 week intervals for up to 8-12 weeks. Study team members will check the patient's medical record for indication of infection or adverse events at each follow-up visit. If no follow up is reported after three months, study staff will conduct a phone interview to collect this data.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients ages 0-17 years old
* Skeletally immature patients, as confirmed by xray imaging evaluated by an orthopaedic surgeon
* Patient as sustained a grade 1 or 2 open fracture within 24 hours of presentation
* Physician plans to manage the fracture non-operatively

Exclusion Criteria:

* Patients 18 years or older
* Skeletally mature patients, as as confirmed by xray imaging evaluated by an orthopaedic surgeon
* Patients with grade 3 open fractures
* Gross contamination of the fracture
* Fracture requires surgery
* Immunocompromised patients
* Allergies to cephalosporins
* Severe penicillin allergy
* non-English speaking patients &/or guardian

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2033-09 (Estimated); Study Completion 2034-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with an infection at the fracture site. | Up to 3 months following injury.
  Participants will be monitored for infection at follow-up appointments and/or through follow-up phone contact.

SECONDARY OUTCOMES:
Drug adverse events | Up to 3 months following injury.
  Any adverse side effects resulting from antibiotics administered.

CONTACTS AND LOCATIONS:
Overall Officials: Sivashanmugam Raju, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States